CLINICAL TRIAL: NCT06916871
Title: Optimizing Care for Diabetic Patients in Hospitalized Rehabilitation Through Structured Education.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Principal Investigator, Helena Cassol, Principal Investigator, Centre Hospitalier Universitaire de Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-416
Record Dates: First submitted 2025-02-11; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus Self Management Education
Keywords: optimisation; autonomie; diabète; réadaptation; éducation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Awareness (Active Comparator): The control group will benefit from awareness. Doctors and nursing staff will transmit information in a linear manner, i.e. explain, possibly argue and answer the patient's questions on topics such as interpreting blood sugar levels, explaining treatment, good practices in terms of diet, physical activity, etc. at the patient's bedside in an unstructured manner based on interactions between patient and caregivers. There is therefore no standard frequency, number of specific sessions, or topics addressed systematically.
  Interventions: Other: The control group will benefit from awareness
- Education (Experimental): The experimental group will benefit from structured education which will be carried out by the diabetes nurse at a rate of 3 sessions for patients on oral anti-diabetics and 5 sessions for patients on insulin.
  Interventions: Other: The experimental group will benefit from structured education which will be carried out by the diabetes nurse

INTERVENTIONS:
Other: The control group will benefit from awareness — During hospitalization in rehabilitation, doctors and nursing staff will transmit information in a linear manner, i.e. explain, possibly argue and answer the patient's questions on topics such as interpreting blood sugar levels, explaining treatment, good practices in terms of diet, physical activity, etc. at the patient's bedside in an unstructured manner based on interactions between patient and caregivers. There is therefore no standard frequency, number of specific sessions, or topics addressed systematically.
  Arms: Awareness
Other: The experimental group will benefit from structured education which will be carried out by the diabetes nurse — During hospitalization in rehabilitation, the experimental group will benefit from structured education which will be carried out by the diabetes nurse at a rate of 3 sessions for patients on oral anti-diabetics and 5 sessions for patients on insulin.
  Arms: Education

SUMMARY:
A large number of patients at the Neurological and Functional Rehabilitation Centre of the University Hospital of Liège have associated pathologies, including diabetes. These patients may have diabetes-related complications that require recurrent hospitalizations in an acute structure or in rehabilitation. One of the ways to limit complications is to set up patient education.

1. Objectives

   * To compare the impact of management through formal education with that of awareness.
   * To evaluate the impact on knowledge of structured education.
   * To evaluate the impact of structured education on the quality of life experienced by diabetic patients.
   * Identify the patient's level of satisfaction with the education sessions.
   * To evaluate the impact of structured education on the biological improvement of glycated hemoglobin.
   * To evaluate the impact of structured education on diabetes-related complications.
2. Working Hypothesis The implementation of structured diabetes education allows "patients to acquire, or maintain, the skills they need to manage their lives as well as possible despite the constraints of chronic disease... ".
3. Study population All diabetic patients hospitalized in all care units.
4. Collection tools and techniques Collection tools

1. "Diabetes Knowledge Questionnaire". 2. SF-36 Health Questionnaire. 3. Satisfaction questionnaire for structured sessions on diabetes. 4. Questionnaire to identify complications and/or re-hospitalizations after your stay in rehabilitation.

Collection technology At admission (D+1)

* Validation of inclusion and exclusion criteria.
* Submission and distribution of the information and consent form.
* Obtaining informed consent from the patient.
* Distribution of collection tools 1 and 2 (collection on D+2).
* Control of glycated hemoglobin. At the end of hospitalization (D-2)
* Distribution of collection tools 1, 2 and 3 on D-2 before the release (collection on D-1).
* Control of glycated hemoglobin. 3 months after the end of hospitalization
* Sending collection tools 1, 2 and 4 by post. The patient will be invited to complete them and return them by post.
* The patient will be invited to take a blood test for glycated hemoglobin.

DETAILED DESCRIPTION:
Introduction The World Health Organization (WHO) defines diabetes as "a chronic disease that occurs when the pancreas does not produce enough insulin, or when the body is unable to use the insulin it produces effectively.

Type 1 diabetes (formerly called insulin-dependent or juvenile diabetes) is characterized by insufficient insulin production, which must be administered daily. In 2017, 9 million people had type 1 diabetes, most of them living in high-income countries. The cause of type 1 diabetes is not known, and it is not currently known how to prevent it.

Type 2 diabetes changes the way the body uses sugar (glucose) for energy. It prevents the body from using insulin properly, which can lead to high blood sugar levels if left untreated. Over time, type 2 diabetes can cause serious damage, especially to nerves and blood vessels. Type 2 diabetes can often be prevented. Factors that contribute to the development of type 2 diabetes include being overweight, not getting enough exercise, and having a genetic predisposition.

One of the most important ways to treat diabetes is to maintain a healthy lifestyle.

Some people with type 2 diabetes will need to take medication to control their blood sugar. This may include injected insulin or other medications, including: metformin, sulfonylureas, sodium-glucose cotransporter-2 inhibitors (SGLT-2 inhibitors). " According to the International Diabetes Federation (IDF), "The facts and figures about diabetes demonstrate the growing global burden it places on individuals, families, and countries. The IDF Diabetes Atlas (2021) indicates that 10.5% of the adult population (20-79 years) have diabetes and nearly half of them are unaware that they are living with the condition.

By 2045, IDF projections show that one in eight adults, or approximately 783 million people, will be living with diabetes, representing an increase of 46%.

More than 90% of people with diabetes have type 2 diabetes, which is due to socioeconomic, demographic, environmental and genetic factors. The main factors contributing to the increase in type 2 diabetes are:

* Urbanization.
* Ageing population.
* Decreased levels of physical activity.
* Increased prevalence of overweight and obesity. However, it is possible to reduce the impact of diabetes by taking preventive measures for type 2 diabetes and providing early diagnosis and appropriate care for all types of diabetes. These measures can help people with diabetes avoid or delay complications. " In Belgium in 2021, 6.8% of the Belgian population suffered from diabetes, which represents 798,912 people. 1/3 of people are not diagnosed with diabetes, which brings the prevalence of diabetes in Belgium to 10% (i.e. more than 1 million people).

Effective management of diabetic patients is therefore a real challenge and is of paramount importance at a time when government budgetary constraints are increasingly severe. The transfer of skills, the financing law and the new method of financing institutions have considerably impacted the financial resources of our hospitals.

How can it be done better with less? How can hospitalizations that are costly for society and their duration be limited within the framework of limited hospital funding?

1. Problem A large number of patients at the Neurological and Functional Rehabilitation Center (CNRF) have associated pathologies, particularly diabetes. These patients may have complications related to diabetes that require recurring hospitalizations in an acute structure or in rehabilitation. One way to limit complications is to implement patient education.

"Patient education consists of nursing care aimed at facilitating the learning of knowledge, know-how and interpersonal skills in order to achieve a change in behavior in the patient, their family or a significant person." Before the implementation of this project, patient education consisted of awareness-raising according to the definition of the 2011 Minimum Hospital Summary Nursing Data Scoring Manual (DI-RHM) "Set of educational activities carried out with the aim of raising awareness, informing or enabling the acquisition of certain knowledge, abilities or skills with a view to regaining autonomy: information on the disease process, education in the management of prescribed medication, etc. These activities concern the patient, their family or any other person

ELIGIBILITY:
Inclusion Criteria:

* Patient having given written consent.
* Diagnosis of diabetes notified in medical file.
* Be at least 18 years old.
* Be able to communicate orally and in writing.
* Have a sufficient understanding of the French language.

Exclusion Criteria:

* Presence of cognitive disorder, confusion, spatio-temporal disorientation noted in the nursing and/or medical file.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-07 (Estimated); Primary Completion 2027-04-07 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Diabete Knowledge Questionnaire. | From the day after the first day of hospitalization in rehabilitation to 3 months after the end of hospitalization.
  The DKQ consists of 15 multiple-choice questions relating to the minimum knowledge about diabetes. Fourteen of the fifteen questions concern type 1 and type 2 diabetes. Question 15 relates only to type 1 diabetes. Demographic data, such as age, gender, duration of diabetes, as well as type of drug treatment, are collected by an additional 16th question consisting of nine items.
  A score of 0 to 1 is assigned to each of the answers to the questions; For some questions, several answers must be checked. A score of 0 is assigned for an incorrect answer, 1 for a correct answer, and 0.5 for "unsure". For participants with type 2 diabetes who are not taking medication, the total possible score is a maximum of 26. It is 28 for people who take anti-diabetic medications. For participants with type 1 diabetes, the maximum possible score is 32.
Quality of life felt. | From the day after the first day of hospitalization in rehabilitation to 3 months after the end of hospitalization.
  The SF-36 short-form questionnaire is used to obtain a generic measure of perceptual health status. Each question is scored with a Lickert with a minimum value of 0 and a maximum value of 100. The lowest values indicate a poorer perceived quality of life and the higher values indicate a better quality of life.

SECONDARY OUTCOMES:
Patient's level of satisfaction. | Two days before the end of hospitalization.
  Patient's level of satisfaction with the structured education program is rated on a scale from 0 (worst/lowest satisfaction status) to 10 (highest satisfaction status).
Improvement of glycated hemoglobin. | From the day after the first day of hospitalization in rehabilitation to 3 months after the end of hospitalization.
  A significant decrease (p < 0.05) in the patient's glycated hemoglobin value is expected.
Diabetes-related complications. | 3 months after the end of hospitalization.
  Follow-up of diabetes-related complications: number of consultations with the general practitioner, number of consultations with the diabetic nurse and number of hospitalizations.

CONTACTS AND LOCATIONS:
Overall Officials: Théodora Giagoultsis, Head nurse, Principal Investigator — Centre Hospitalier Universitaire de Liege; Justine Slomian, scientist, Principal Investigator — Centre Hospitalier Universitaire de Liege; Nadia Jaajouai, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (1):
- Centre Hospitalier Universitaire de Liège, site Centre Neurologique et de Réadaptation Fonctionnelle, Tinlot, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No